CLINICAL TRIAL: NCT00704509
Title: A Multinational, Randomised, Double-Blind, Fixed-Dose, Bifeprunox Study Combining a 12-Week Placebo-Controlled, Quetiapine-Referenced Phase With a 12-Month Quetiapine-Controlled Phase in Patients With Schizophrenia
Brief Title: Efficacy of Bifeprunox in Patients With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis showed inadequate efficacy of bifeprunox
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11916A; 2007-001098-27 (EudraCT Number)
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; Bifeprunox
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bifeprunox (Experimental)
  Interventions: Drug: Bifeprunox
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Quetiapine (Active Comparator)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Bifeprunox — 20 mg daily, encapsulated tablets, orally, 12 months
  Other Names: DU 127090
  Arms: Bifeprunox
Drug: Placebo — Encapsulated tablets, orally, 12 weeks
  Arms: Placebo
Drug: Quetiapine — 600 mg daily, encapsulated tablets, orally, 12 months
  Other Names: Seroquel
  Arms: Quetiapine

SUMMARY:
The primary purpose of the study is to evaluate the efficacy of bifeprunox in the maintenance phase of schizophrenia compared to placebo.

DETAILED DESCRIPTION:
Schizophrenia is a serious and disabling mental disorder that affects approximately 1% of the world's population. There are a number of antipsychotic drugs in use but none is ideal, in particular because their safety profile is complex and their effectiveness is limited. In particular, after having overcome acute exacerbations many patients continue to experience significant symptoms that prevent an adequate functioning. In the current study, patients suffering from schizophrenia and currently in a post-acute maintenance phase of the disease will be included. Non-treatment resistant patients will be included in the study, since they have partially responded to their current antipsychotic treatment but still have clinically significant symptoms and/or impairment of functioning in their daily life. The study is a 12-month study with an initial 12-week placebo-controlled, quetiapine-referenced phase. After this initial 12-week phase, the patients allocated to placebo will be switched to bifeprunox. In the final non-inferiority analysis of the 12-month data, the results from this study will be combined with the data from a similar study (11915A).

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria

* The subject has a primary diagnosis of schizophrenia
* The subject experiences clinically significant symptoms
* The subject's medication remained stable for 8 weeks prior to screening
* The subject is currently in the post-acute maintenance phase of his/her disease

Exclusion Criteria:

Main exclusion criteria

* The subject is at significant risk of suicide
* The subject is treatment resistant
* The subject has experienced an acute exacerbation within 8 weeks prior screening
* The subject is unlikely to comply with the protocol
* The subject has a current diagnosis or a history of substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The difference in change from baseline to the 12-week time point between bifeprunox and placebo using the Positive and Negative Syndrome Scale (PANSS). | 12 weeks

SECONDARY OUTCOMES:
The difference in PANSS score at the 12-month time point between bifeprunox and quetiapine. Also, responder rate, time to response/withdrawal, global clinical assessments (CGI), assessment of depressive symptoms (CDSS) and health economic assessments. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (45):
- India (10):
  - IN008, Ahmedabad
  - IN011, Ahmedabad
  - IN009, Aurangabad
  - IN003, Bangalore
  - IN006, Chennai
  - IN007, Kanpur
  - IN002, Lucknow
  - IN001, Mangalore
  - IN010, Varanasi
  - IN005, Visakhapatnam
- Indonesia (3):
  - ID002, Bangli
  - ID001, Jakarta
  - ID003, Kabupaten Bandung
- Malaysia (4):
  - MY005, Johor Bahru
  - MY001, Kuala Lumpur
  - MY004, Kuala Lumpur
  - MY003, Perak
- Philippines (5):
  - PH004, Cebu City
  - PH001, Mandaluyong
  - PH002, Manila
  - PH003, Pasig
  - PH005, Quezon City
- Poland (8):
  - PL005, Choroszcz
  - PL007, Kutno
  - PL002, Leszno
  - PL004, Lodz
  - PL003, Lublin
  - PL008, Skorzewo
  - PL006, Swicie n/Wisla
  - PL001, Torun
- South Korea (6):
  - KR004, Busan
  - KR008, Gyeongnam
  - KR005, Pusan
  - KR006, Seoul
  - KR001, Seoul
  - KR007, South Korea
- Ukraine (9):
  - UA008, Dnipropetrovsk
  - UA009, Donetsk
  - UA006, Kharkiv
  - UA003, Kyiv
  - UA004, Lviv
  - UA011, Odesa
  - UA005, Poltava
  - UA007, Stepanovka, Kherson
  - UA010, Vinnitsa

REFERENCES:
- [Derived] Ceraso A, Lin JJ, Schneider-Thoma J, Siafis S, Tardy M, Komossa K, Heres S, Kissling W, Davis JM, Leucht S. Maintenance treatment with antipsychotic drugs for schizophrenia. Cochrane Database Syst Rev. 2020 Aug 11;8(8):CD008016. doi: 10.1002/14651858.CD008016.pub3. PMID 32840872